CLINICAL TRIAL: NCT05111990
Title: The Influence of Maternal Health on Human Breast Milk Composition With Potential Downstream Effects on Infant Metabolism and Gut Colonization
Brief Title: Human Milk and Its Effect on Infant's Metabolism and Infant Gut Microbiome
Acronym: MAINHEALTH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); Arla Foods (Industry); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-296-18
Record Dates: First submitted 2021-09-24; First posted 2021-11-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Milk Collection; Human Milk/Breastfeeding; Human Milk Microbiome; Infant Gut Microbiome
Keywords: milk metabolites, multi-omics, gut microbiome
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample (mother, Gestational age (GA) week 20-24) Vaginal swap (Copan Eswab; mother at birth) Rectum swap (Copan Eswab; mother at birth) Breast milk (3, 30, 60, 90 days postpartum) Urine (infant; 30, 60, 90 days postpartum) Feces (infant; 30, 60, 90 days and 1, 2, 3, 4, and 5 years postpartum) Saliva (Copan Eswab; infant 30 days postpartum) Breast skin (Copan Eswab; mother 30 days postpartum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Maternal pre-gestational BMI 18.5<25
- Maternal pre-gestational BMI 25<30
- Maternal pre-gestational BMI >30

SUMMARY:
This protocol explains the MAINHEALTH cohort. The study examine the influence of maternal health parameters on human breast milk composition and integrates milk phenotype with infant metabolism and infant gut microbial content and metabolism.

DETAILED DESCRIPTION:
The birth of a living human being is the result of an approximately nine-month pregnancy in which the developing foetus has taken exactly the building blocks necessary to grow and develop from its mother. However, growth and development continues in multiple dimensions at an increasing pace after birth. The nutrition in the first 1,000 days from conception to the child's 2nd birthday plays a pivotal role in shaping the future health of the child. Yet, little is known of how breast milk components vary due to maternal factors or of the biological mechanisms behind the beneficial actions of many breast milk nutrients. The investigators propose to overcome these obstacles by combining specialties to give a more complete account of what breast milk is (major and minor milk constituents and microbiota), how it affects the infants directly or indirectly through breast milk-gut microbiome interactions and by which mechanisms. In this study longitudinal samples from 200 mother-infant dyads during the first year of life across three groups of pregestational maternal BMI; normal weight (BMI 18.5-24.99), overweight (BMI 25-30), and obese (BMI >30) are collected. The samples give a comprehensive record of what the infant has ingested (milk samples) and how the infant and infant gut microbiome responds to this (infant urine and feces). Maternal diet in pregnancy and at milk sample deliveries are recorded through a 24h online food recall and diary system. Maternal health attributes will, besides BMI, be analysed through clinical blood biochemistry parameters. Follow-up samples and infant dietary intake as the infant grows allow investigating how early life diet shaped infant growth and gut colonization more long term. The investigators have formed an experienced team of scientists within metabolomics, microbiology and medicine, holding leading positions within their respective fields in Denmark. The novelty in the study is the interdisciplinarity, unique study design and the emphasis to integrate a number of dynamic measurements thereby offering the ability to identify the factors in breast milk affecting infant metabolism and gut colonization. Knowing this enable the optimization of infant formula.

The research questions asked in this project are three-fold.

* First, the investigators want to determine the variability of breast milk nutrients by application of multi-omics (metabolomics, proteomics and glycomics). The production of human breast milk has a high maternal metabolic cost. Thus, hypothesis is that maternal health attributes (metabolic dysfunction or obesity) influence which breast milk nutrients are made available to the infant.
* Second, the investigators want to establish the microbiome of breast milk. Maternal obesity can lead to an apparent gut microbial ecology and increases the risk of obesity for the child. Thus, the hypothesis is that maternal obesity confers distinct microorganisms to the infant.
* Third, the investigators want to identify biological mechanisms for how breast milk nutrients are metabolised in the infants. Infants exclusively breast-feeding offer total compliance. Thus, the hypothesis is that by deconstructing breast milk components and markers of infant metabolism through comprehensive analysis of infant urine and feces, bioactivity of breast milk nutrients can be elucidated.

ELIGIBILITY:
Inclusion Criteria related to mother:

* Residing in Aarhus area
* Above 18 years of age
* BMI above 18.5 kg/m2
* Intention to breastfeed the first four to six months following birth
* Be able to communicate in Danish

Exclusion Criteria related to mother:

* Smoking
* Multiple gestation
* Suffering from the following chronic diseases that demands medical treatment: diabetes mellitus, celiac disease, inflammatory bowel disease (Chrohn's disease or ulcerosa colitis)
* Taking medicaments for irritable bowel syndrome
* Taking medicine for metabolic disorders
* Taking medicine for psychological disorders
* Have had gastric bypass surgery
* Planned caesarean section
* Received antibiotics after week 12 in their pregnancy
* Utilizing significant amount of infant formula following birth

Inclusion Criteria related to infant:

* Infants born after gestational age 37 weeks
* Infants with a birth weight between 2500 g and 5000 g

Exclusion Criteria related to infant:

• Inborn errors of metabolism

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residence in Aarhus area is necessary and Aarhus University Hospital has to be the place of giving birth. This is due to samples being collected by midwifes during labor and when study personnel collect samples in study participants' homes.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Metabolite profile of human milk | Birth to 3 months
  Human milk metabolites by Nuclear Magnetic Resonance (NMR) spectroscopy. Data will be analysed as absolute concentrations of milk metabolites; how milk metabolite profiles are related to mother's blood chemistry, milk microbial profiles, milk oligosaccharides, infant urine metabolome, and infant fecal microbiomes will be explored using multivariate analyses.

SECONDARY OUTCOMES:
Metabolite profile of human milk by Liquid Chromatography-Mass Spectrometry (LC-MS) analysis | Birth to 3 months
  Human milk metabolites by LC-MS-based metabolomics. Data will be analysed as absolute concentrations of milk metabolites; how milk metabolite profiles are related to milk microbial profiles, milk oligosaccharides, infant urine metabolome, and infant fecal microbiomes will be explored using multivariate analyses.
Milk proteome profile | Birth to 3 months
  Human milk proteome by LC-MS-based, bottom-up proteomics. Data will be analysed as relative abundances of milk proteins.
Milk protein post-translational modification (PTM) profile | Birth to 3 months
  Post-translational modifications of human milk proteins is analysed by LC-MS-based and 2D- gel-based proteomics. Data will be analysed as relative abundances of milk protein PTMs.
Milk glycome profile | Birth to 3 months
  Human milk glycome by LC-MS-based glycomics. Data will be analysed as relative abundances of milk glycans.
Microbial structure of human milk | Birth to 3 months
  Human milk microbiome by nanopore sequencing. Data will be analysed as relative abundances of bacteria from phylum to genus levels.
Microbial structure of infant feces | Birth to 5 years of age
  Infant fecal microbiome by nanopore sequencing. Data will be analysed as relative abundances of bacteria from phylum to genus levels.
Microbial structure of infant oral cavity | 30 days postpartum
  Oral cavity microbiome by nanopore sequencing. Data will be analysed as relative abundances of bacteria from phylum to genus levels.
Microbial structure of mother's skin microbiome | 30 days postpartum
  Skin microbiome by nanopore sequencing. Data will be analysed as relative abundances of bacteria from phylum to genus levels.
Metabolite profile of infant fecal material | Birth to 5 years of age
  Infant fecal metabolome by NMR-based metabolomics. Data will be analysed as absolute concentrations of fecal metabolites
Infant metabolism investigated by infant urine metabolomics | Birth to 3 months of age
  Infant urine metabolome by NMR-based metabolomics. Data will be analysed as absolute concentrations of urine metabolites
Microbial structure of maternal vagina and rectum to investigate vertical transmission of bacteria to infant during birth | During birth
  Vertical transmission of microbiome from mother to infant. Vaginal and rectal microbiome by nanopore sequencing. Data will be analysed as relative abundances of bacteria from phylum to genus levels.
Mother's 24-h dietary recall (myfood24) | During pregnancy (Gestational age 30), 30, 60, and 90 days postpartum. In each case two times within a week (one weekday and one weekend day).
  Aggregated nutrient intake data (e.g. proteins, vitamins, fibers, omega-3-fatty acids)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik K Sundekilde, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- [Background] Overgaard Poulsen K, Astono J, Jakobsen RR, Uldbjerg N, Fuglsang J, Nielsen DS, Sundekilde UK. Influence of maternal body mass index on human milk composition and associations to infant metabolism and gut colonisation: MAINHEALTH - a study protocol for an observational birth cohort. BMJ Open. 2022 Nov 2;12(11):e059552. doi: 10.1136/bmjopen-2021-059552. PMID 36323479